CLINICAL TRIAL: NCT01047423
Title: Targeting Microvascular Dysfunction in Young Hypertensive Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Gary E McVeigh, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-011638-90
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Hypertension
Keywords: Hypertension endothelial dysfunction statin prevention
MeSH Terms: conditions — Hypertension | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Experimental): 40mg Simvastatin once daily for 12 weeks followed by 4 week washout period followed by placebo for 12 weeks
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Placebo for 12 weeks followed by 4 week washout period followed by 40mg Simvastatin once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 40mg encapsulated once daily for 12 weeks
  Arms: Simvastatin
Drug: Placebo — Encapsulated oral once daily for 12 weeks
  Arms: Placebo

SUMMARY:
Cholesterol and blood pressure lowering tablets have been shown to be of benefit in patients with established high blood pressure. High blood pressure is a very common medical condition that can lead to vascular complications i.e. problems with the blood vessels in the body. One way of detecting early changes in these blood vessels as a result of high blood pressure is to measure their compliance/flexibility with a noninvasive technique known as ultrasound and with a simple blood test. The investigators are trying to establish whether these early changes in blood vessels can be significantly improved by the use of both a cholesterol and blood pressure lowering tablet at an earlier stage than is currently advised. The investigators hope that the early combination of these tablets will prove more effective than the use of a blood pressure lowering tablet by itself and therefore possibly reduce the risk of long term complications developing.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, all of the following criteria must be met:

  * All patients must have a diagnosis of essential hypertension with off treatment systolic pressure >140 mmHg and/or diastolic pressure >90 mmHg, measured at rest in the seated position on at least two separate occasions, at least 2 weeks apart.
  * Patients will be < 50 years for men and < 60 years for women.
  * Female patients of childbearing potential must be using a medically accepted means of contraception (that is, interuterine device, oral contraceptive, implant, DepoProvera or barrier devices). Female patients of childbearing age will be screened with a pregnancy test.
  * Patients will be typically already on antihypertensive therapy.
  * Patients must have a level of understanding sufficient to complete all tests and examinations required by the protocol and are able to understand and give informed consent.

Exclusion Criteria:

* Patients will be excluded from the study if they meet any of the following criteria:

  * A history of diabetes mellitus, coronary artery or cerebrovascular disease, hypertensive retinopathy, hypertensive nephropathy, left ventricular hypertrophy or hyperlipidaemia warranting treatment as defined by the latest NICE guidelines which recommend an age based treatment strategy rather than one driven purely by lipid levels in isolation.
  * Abnormal baseline liver function (defined as AST or ALT > 3 times upper limit of normal), raised baseline creatinine kinase (CK) (defined as CK > 200 mmol/L), severe renal impairment (defined as estimated glomerular filtration rate (eGFR) < 30 mls/minute) or previous adverse event relating to either an ARB or statin in the past.
  * Female patients will be excluded if they are pregnant, intend to be pregnant or are lactating. Female patients of childbearing age will be screened with a pregnancy test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
To demonstrate a significant difference in flow-mediated dilatation of the brachial artery and microvasculature between groups. | 0, 3, 4 and 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary E McVeigh, FRCP PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Belfast health and social care trust, Belfast, United Kingdom

REFERENCES:
- [Derived] Bleakley C, McCann A, McClenaghan V, Hamilton PK, Millar A, Pumb R, Harbinson M, McVeigh GE. Ultrasound entropy may be a new non-invasive measure of pre-clinical vascular damage in young hypertensive patients. Cardiovasc Ultrasound. 2015 Mar 20;13:12. doi: 10.1186/s12947-015-0006-7. PMID 25888961